CLINICAL TRIAL: NCT05196204
Title: Trunk Task-oriented Training Combined With Functional Electrical Stimulation to Improve Functional Independence, Postural Control and Neuroplasticity in Spinal Cord Injured Individuals
Brief Title: Trunk Task-oriented Training Combined With Functional Electrical Stimulation in Spinal Cord Injured Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Collaborators: Mitacs (Industry); Neuro-Concept Inc. (Unknown)
Responsible Party: Principal Investigator, Dorothy Barthélemy, Associate professor and researcher, Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRIR-1497-1020
Record Dates: First submitted 2021-09-01; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Spinal Cord Injuries
Keywords: Trunk task-oriented training; Corticospinal tract; Functional electrical stimulation; Functional independence; Trunk motor control
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trunk-oriented task combined with functional electrical stimulation training group (Experimental): This group will be formed with participants with spinal cord injury. This group will perform 12 weeks of trunk-oriented task training combined with functional electrical stimulation.
  Interventions: Other: Trunk-oriented task training combined with functional electrical stimulation
- Trunk-oriented task training group (Active Comparator): This group will be formed with participants with spinal cord injury. This group will perform 12 weeks of trunk-oriented task training.
  Interventions: Other: Trunk-oriented task training alone
- Control group (No Intervention): Healthy participants will be recruited based on the age and sex of the participants with spinal cord injury to realize clinical, biomechanical and cortical evaluations

INTERVENTIONS:
Other: Trunk-oriented task training combined with functional electrical stimulation — Training will consist to perform one hour of trunk task-oriented training combined with functional electrical stimulation (FES/T-TOT) specific for muscle strength and motor control. All training will be done seated without support with knees and hips flexed to 90 degrees. FES will be combined with functional and non-functional tasks to work functionality and muscle strengthening. Each training session will consist on the fulfilment of two functional tasks (as reaching) and two non-functional tasks (as push-up movement) from a battery of postural control exercises.
  Arms: Trunk-oriented task combined with functional electrical stimulation training group
Other: Trunk-oriented task training alone — The SCI participants who will perform T-TOT training alone will have to perform the same exercises as explained in the previous section (two functional tasks and two non-functional tasks) but they will not receive any functional electrical stimulation.
  Training will consist to perform one hour of trunk task-oriented training (T-TOT) specific for muscle strength and motor control. All training will be done seated without support with knees and hips flexed to 90 degrees. Each training session will consist on the fulfilment of two functional tasks (as reaching) and two non-functional tasks (as push-up movement) from a battery of postural control exercises.
  Arms: Trunk-oriented task training group

SUMMARY:
The objectives of the study are to evaluate trunk task-oriented training combined with function electrical stimulation (FES/T-TOT) efficacy on sitting balance and functional independence, and to understand the mechanisms of neuroplasticity that would improve functional independence following FES/T-TOT in individuals with spinal cord injury.

DETAILED DESCRIPTION:
After obtaining their consent, participants will undertake evaluations at different times:

1. Assessment 3 weeks prior to training
2. Assessment 1 week prior to training
3. Training over 12 weeks
4. Assessment 1 week after training
5. Assessment 1 month after training (follow-up)

Each assessment will be divided in 2 sessions and data will be collected over 2 days, at one session per day. The assessment will consist of:

* Session 1 (at Neuro-Concept clinic) will include presentation of the study and the obtention of written consent, clinical (modified Reaching test and muscle strength), quality of life and functional independence assessments.
* Session 2 (at IURDPM in Dr. Barthélemy's laboratory) will include postural control, corticospinal and cortical assessments.

After the initial assessment, the participants with spinal cord injury will realize 36 sessions of trunk task-oriented training alone or combined with function electrical stimulation (3 times a week for 12 weeks).

ELIGIBILITY:
FOR PARTICIPANTS WITH SPINAL CORD INJURY

Inclusion Criteria:

* Level of spinal cord lesion between C6/C7 and T10
* At least, 6 months post-injury
* Be considered as AIS A, B, C or D
* Be able to sit without support for 15 seconds
* Be able to provide informed consent in English or in French

Exclusion Criteria:

* To have cognitive deficits
* To wear a corset
* To have personal or family history of epilepsy
* To have suffered moderate or severe traumatic brain injury
* To have cochlear implant

FOR CONTROL PARTICIPANTS

Exclusion Criteria:

* To have orthopedics problems
* To have cognitive deficits
* To have neurological problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Change in Function in Sitting Test | Before and after the 12-week trainings and 1-month follow-up
  This test evaluates the sitting balance via 14 everyday functional activities rated from 0 to 4 according to the reactions of the participants.
Change in modified Functional Reach Test | Before and after the 12-week trainings and every 4-weeks during the training period
  This test evaluates the ability for each participant to realize a lateral and anterior trunk flexion in order to observe the maximum distance reached.

SECONDARY OUTCOMES:
Change in EMG activation pattern of electromyographic activity of muscles in the trunk | Before and after the 12-week trainings and 1-month follow-up
  during reaching and pointing tasks
Change in the center of pressure excursion | Before and after the 12-week trainings and 1-month follow-up
  during reaching and pointing tasks
Modification of the excitability of the reticulospinal pathway using the acoustic startle response | Before and after the 12-week trainings and 1-month follow-up
  A tone will be triggered just before the reaching movement. The EMG responses of trunk muscles will be analyzed.
Modification of the excitability of the vestibulospinal pathway using galvanic vestibular stimulation | Before and after the 12-week trainings and 1-month follow-up
  Vestibular responses induced by GVS will be identified in the trunk muscles

OTHER OUTCOMES:
Physical Activity Recall Assessment for People with Spinal Cord Injury (questionnaire) | Before and after the 12-week trainings
  This interview will capture all physical activity information over the previous 3 days. Eight periods of day will be screened (morning routine, breakfast, morning, lunch, afternoon, dinner, evening, evening routine). This test allows us to verify if the intensity of daily physical activity of each participant will be constant during the intervention.
Change in quality of life using World Health Organization Quality of Life with disabilities module (WHOQOL-BREF) | Before and after the 12-week trainings and 1-month follow-up
  This questionnaire consists in 39 questions about participant feelings.
Change in quality of life using Short-Form 36 questionnaire | Before and after the 12-week trainings and 1-month follow-up
  The questionnaire consists in 36 questions about 8 domains: physical functioning, role functioning-physical, bodily pain, general health, vitality, social functioning, role functioning-emotional and mental health
Change in the Quality of life index | Before and after the 12-week trainings and 1-month follow-up
  This questionnaire consists in 37 questions about 4 domains: health and functioning, psychological/spiritual, social and economic, and family.
Change in functional independence using Spinal Cord Independence Measure questionnaire | Before and after the 12-week trainings and 1-month follow-up
  This questionnaire consists in evaluation of self-care, respiration and sphincter management, and a participant's mobility abilities.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Neuro-Concept Inc, Montreal, Quebec
  - Neuromobility lab, Montreal, Quebec